CLINICAL TRIAL: NCT01508572
Title: Validation of Uptake of a VEGF-targeted Optical Fluorescent Imaging Tracer in Surgical Specimens of Breast Cancer and Application of Pre- and Intra-operative Human Molecular Fluorescence Imaging Techniques. A Multicenter Feasibility Study
Brief Title: VEGF-targeted Fluorescent Tracer Imaging in Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Principal Investigator, G.M. van Dam, Prof Dr, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCG/UMCU_01; 2011-003083-75 (EudraCT Number)
Record Dates: First submitted 2011-12-22; First posted 2012-01-12 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; VEGF; optical imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab-IRDye800CW (Experimental): In this two stage, non-randomized, non-blinded, prospective, multicenter feasibility study, bevacizumab-IRDye800CW will be administered to a total of 20 patients with proven breast cancer.
  Interventions: Drug: bevacizumab-IRDye800CW

INTERVENTIONS:
Drug: bevacizumab-IRDye800CW — In this two stage, non-randomized, non-blinded, prospective, multicenter feasibility study, bevacizumab-IRDye800CW will be administered to a total of 20 patients with proven breast cancer.
  Other Names: Fluorescence tracer imaging; Beva-800CW; Bevacizumab-800CW

SUMMARY:
The purpose of this study is to determine the uptake, (semi-)quantification and localization of the VEGF targeting fluorescent tracer bevacizumab-IDRye800CW in breast cancer tissue, surrounding healthy tissue, tumor margins and lymph nodes. This is measured in surgical specimens after a single intravenous administration of 4,5 bevacizumab-IDRye800CW, using fluorescence microscopy and macroscopy techniques. Also the safety of bevacizumab-IDRye800CW is assessed. Another purpose is to assess the abilities of three different fluorescent signal detection systems to detect the fluorescent signal pre- and intra-operatively.

DETAILED DESCRIPTION:
There is a need for better visualization of presence and extent of breast cancer to improve breast cancer management. Molecular imaging of breast cancer associated targets is a promising method to improve visualization. Vascular endothelial growth factor (VEGF) has proven to be a valid target for molecular imaging with radioactive labeled tracers. However in view of radiation safety, infrastructure, costs and stability, fluorescent labeling of bevacizumab (a VEGF targeting humanized monoclonal antibody) has potential advantages over radioactive labeling. Therefore recently the near-infrared fluorescent tracer bevacizumab-IRDye 800CW has been developed. In mice the fluorescent signal was clearly present in tumor tissue and could be visualized intra-operatively. The tracer was also approved for administration to patients in a microdose (tracer dose).

In this prospective multicenter feasibility study the new tracer bevacizumab-IRDye 800CW will be administered to a maximum of 30 patients with proven breast cancer 3 days before surgery. Part of the surgical specimen will after surgery extensively be investigated by macroscopy and microscopy to determine the uptake of the tracer in tumor tissue, surrounding normal tissue and lymph nodes. To detect the tracer before surgery, two different pre-operative imaging methods are used: MSOT (in the UMCG en FDOT in the UMCU. During surgery the intra-operative MFRI camera is available at both centers to detect the fluorescent signal.

The study consists of a total of five study procedure related patient visits.

1. During a screening visit, eligibility will be evaluated and patient characteristics will be collected.
2. During the administration visit, 3 days before surgery, 4.5 mg of bevacizumab-IRDye 800CW will be administered intravenously, followed by 4 hours observation. Also before and 4 hours after tracer injection pre-operative optical imaging will take place (in the UMC Groningen, the hand-held MSOT system will be used and in the UMC Utrecht, the FDOT system will be used) and blood samples are taken.
3. A third visit, approximately 36 hours after tracer administration, another pre-operative optical imaging procedure will take place.
4. At the day of surgery, first a blood sample will be taken and the last pre-operative optical imaging procedure will take place, followed by standard surgery. During surgery, the MFRI camera will be used to detect a fluorescent signal before and after incision an after removal of the tumor. Part of the surgical specimen will after surgery extensively be investigated by macroscopy and microscopy to determine the uptake of the tracer in tumor tissue, surrounding normal tissue and lymph nodes.
5. At an outpatient visit (approximately 10 days after surgery) (visit 5), the last blood sample will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients with proven breast cancer (cytology, histology) who are scheduled to receive operation intervention.
* Tumor size of at least 15 mm diameter according to anatomical imaging data.
* Signed written informed consent.
* Able to comply with the protocol.
* WHO performance score 0-2.

Exclusion Criteria:

* Other invasive malignancy.
* Serious other medical conditions.
* Pregnant or lactating women. (Documentation of a negative pregnancy test must be available for pre-menopausal women with intact reproductive organs and for women less than two years after menopause).
* Prior radiotherapy on the involved area.
* Major surgery within 28 days before the initiation of the study.
* Prior allergic reaction to immunoglobulins or immunoglobulin allergy.
* Prior neo-adjuvant chemotherapy.
* Breast prosthesis in target breast.

UMC Utrecht (FDOT) specific exclusion criteria

* Breast is too big to fit in the biggest cup or is too small to fit in the smallest cup of the FDOT system.
* Non-intact skin at time of the FDOT procedures.
* Breast located skin diseases.
* Piercings or tattoos located on the breast/nipple.
* Contra-indication for MR procedures or claustrophobia.
* Inability to lay prone positioned for the duration of the FDOT procedure (10 minutes) and MR procedure (30 minutes).
* Tumor located close to the chest wall as assessed by breast imaging data.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The uptake of bevacizumab-IRDye800CW in breast cancer tissue, surrounding tissue and lymph nodes in surgical specimens by fluorescence microscopy and macroscopy | After the last patient is included, which is expected to be within one year after the first inclusion
  Outcome measures:
  * The accumulation, tissue distribution, lokalization and (semi) quantification of bevacizumab-IRDye800CW in breast cancer tissue, surrounding tissue and lymph nodes. Measured by macroscopy using MSOT, Odessey and MFRI and by microscopy using fluorescence microscope and Odessey.
  * Correlation of the above to VEGF-levels and other biological parameters.
Occurrence of adverse events as a measure of safety and tolerability of bevacizumab-IRDye800CW | Participants will be observed for the duration of hospital stay, an expected average of 4 hours after tracer injection. In case of adverse events, patients are observed and treated until recovery
  Obtaining information on safety aspects of bevacizumab-IRDye 800CW, side effects, AE, SAE, SUSAR by observing patients after tracer injection and follow up until 14 days after surgery

SECONDARY OUTCOMES:
Detection ability of preoperative optical fluorescence imaging techniques (FDOT; Fluorescence diffuse optical tomography and MSOT; multispectral opto-acoustic imaging) of the fluorescent signal from bevacizumab-IRDye800CW | detection of the tracer is performed at 4h, 36h and 72h after tracer injection.
  * To assess and compare the presence of a fluorescent signal in breast cancer tissue and normal tissue
  * To explore pharmacokinetics and optical imaging time-points by peforming FDOT/MSOT at multiple time points after administration.
  * To correlate the fluorescence signal assessed by FDOT/MSOT with VEGF-levels, other biological parameters and the fluorescent signal assessed in the ex-vivo surgical specimen.
Detection ability of the intra-operative mulitspectral fluorescence reflectance imaging (MFRI) of the fluorescent signal from bevacizumab-IRDye 800CW during surgery | 72 hours after tracter injection, during surgery.
  * To assess and compare the presence of a fluorescent signal in breast cancer tissue and normal tissue by assessing the images made by the MFRI during and after surgery.
  * the fluorescent signal assessed by MFRI will be correlated with VEGF levels in the ex-vivo surgical specimens.
Detection ability of all optical imaging techniques (FDOT, MSOT, MFRI) of the fluorescent signal in surgical specimens ex vivo | after the last patient is operated, which is approximately one year after study start.
  Assessment of the ability of all optical imaging techniques (FDOT, MSOT, MFRI) to detect fluorescent signal in surgical specimens ex vivo by (semi) quantification of the images and to compare images between different techniques and different tissues (surrounding tissue, tumor tissue and lymph nodes)

CONTACTS AND LOCATIONS:
Overall Officials: Go M. van Dam, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands